CLINICAL TRIAL: NCT03311503
Title: Phase I/II Trial of Lentiviral Gene Transfer for SCID-X1 With Low Dose Targeted Busulfan Conditioning
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Williams (Other)
Responsible Party: Sponsor-Investigator, David Williams, Chief Hematology Oncology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00023098
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Severe Combined Immunodeficiency, X Linked; Gene Therapy
Keywords: lentiviral; Gene therapy; busulfan
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: open labeled, multi-center, phase I/II, cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) lentiviral vector G2SCID
  Interventions: Biological: autologous CD34+ cell transduced with G2SCID vector

INTERVENTIONS:
Biological: autologous CD34+ cell transduced with G2SCID vector — single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) lentiviral vector G2SCID

SUMMARY:
This is a phase I/II open label multi-center study in which patients will receive low dose targeted busulfan followed by infusion of autologous CD34+ selected bone marrow or mobilized peripheral blood cells transduced with the G2SCID vector. Subjects will be enrolled over 3 years and be followed for 2 years post-infusion on this protocol, then followed long-term on a separate long-term follow-up protocol.

Enrollment of subjects will be agreed upon by representatives of both sites. Data will be collected uniformly from both sites through an electronic capture system and key laboratory studies will be centralized.

Harvest, cellular manufacturing and infusion will occur at each site using the same SOPs. Key aspects of cellular product characterization will be centralized

DETAILED DESCRIPTION:
This is an open labeled, multi-center, phase I/II, cohort study involving a single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) lentiviral vector G2SCID in up to 10 patients with X-linked SCID (SCID-X1) at Boston Children's Hospital, UCLA Mattel Children's Hospital, Cincinnatti Childrens Hospital Medical Center, Children's Healthcare of Atlanta. Patients will receive transduced cells after low dose targeted busulfan pre-conditioning (n=12).

Enrolled subjects will be followed for 2 years after infusion on this protocol. Required long-term monitoring for a total of 15 years after infusion will be performed on a separate protocol.

Single infusion of autologous CD34+ cells transduced with the SIN lentiviral vector rHIV_IL2RGcoG2SCID (hereafter G2SCID) The primary objective is to measure event free survival and T cell immune reconstitution at 1 year post-infusion

Secondary objectives are to measure overall survival, event-free survival, safety related to the procedure, and clinical and laboratory measures of efficacy including humoral immune reconstitution and gene marking after gene transfer.

Exploratory objectives include: molecular characterization of gene transfer, detailed assessment of biomarkers of T and B cell development and function, assessment of infections, nutritional status, growth and development post gene therapy, assessment of T cell receptor and B cell receptor repertoire by next generation sequencing, correlation of busulfan levels with immune outcome and molecular measurements of gene transfer

ELIGIBILITY:
Inclusion Criteria:

- 1. Diagnosis of SCID-X1 based on immunophenotype and lack of T cell function (proliferation to PHA <10% of the lower limit of normal for the laboratory) AND confirmed by a mutation in IL2RG 2. Lack of an HLA identical (A, B, C, DR, DQ) related donor 3. Age 5 years old or younger 4. Signed informed consent 5. Documentation of willingness to follow up for 15 years post-infusion as currently required by the FDA 6. If the patient has previously undergone allogeneic transplant, lack of donor T cell engraftment must be documented.

7. Age at least 8 weeks by the time of busulfan administration

Exclusion Criteria:

1. Patients with an active, therapy-resistant infection. Infections that are known to be highly morbid in SCID patients will be considered active and therapy-resistant if the infectious agent is repeatedly isolated despite a minimum of 2 weeks of appropriate therapy and is associated with significant organ dysfunction (including but not limited to abnormalities listed below).

   1. Mechanical ventilation including continuous positive airway pressure
   2. Abnormal liver function defined by AST and ALT >10 times the upper range of normal OR Bilirubin >2 mg/dL
   3. Shortening fraction on echocardiogram <25% or ejection fraction <50%
   4. Renal failure defined as glomerular filtration rate <30 ml/min/1.73 m2 or dialysis dependence
2. Uncontrolled seizure disorder
3. Encephalopathy
4. Documented coexistence of any disorder known to affect DNA repair
5. Diagnosis of active malignant disease other than EBV-associated lymphoproliferative disease
6. Patients with evidence of infection with HIV-1
7. Major (life-threatening) congenital anomalies. Examples of "major (life-threatening) congenital anomalies" include, but are not limited to: unrepaired cyanotic heart disease, hypoplastic lungs, anencephaly or other major central nervous system malformations, other severe non-repairable malformations of the gastrointestinal or genitourinary tracts that significantly impair organ function.
8. Other conditions which in the opinion of the P.I. or co-investigators, contra-indicate collection and/or infusion of transduced cells or indicate patient's inability to follow the protocol. These may include for example clinical ineligibility to receive anesthesia, severe deterioriation of clinical condition of the patient after collection of bone marrow but before infusion of transduced cells, or documented refusal or inability of the family to return for scheduled visits. There may be other unforeseen rare circumstances that would result in exclusion of the patient, such as sudden loss of legal guardianship

   -

Ages: 0 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — X linked
Enrollment: 12 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to measure event free survival | 1 year post infusion
  Events will include death, infusion of unmanipulated back-up product for failure of hematopoietic recovery, and allogeneic transplant performed for poor immune reconstitution
T cell reconstitution | 1 year post infusion
  * CD3+ T cell count ≥300 cells/microliter in peripheral blood
  * Gene marking ≥0.1 copies/cell in sorted CD3+ T cells

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Yun Pai, MD, Study Chair — National Institutes of Health (NIH)
Locations (4):
- United States (4):
  - Mattel Children's Hospital - UCLA, Los Angeles, California
  - Emory University/Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Boston Childrens Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided